CLINICAL TRIAL: NCT04045366
Title: Impact of Capillary Leak and Hypoalbuminemia on PK/PD of Anidulafungin and Caspofungin in Critically Ill Patients
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Collaborators: KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S54510
Record Dates: First submitted 2019-06-14; First posted 2019-08-05 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-07

CONDITIONS: Critically Ill Patients
Keywords: Pharmacokinetics; Echinocandins; Critically ill patients
MeSH Terms: interventions — Specimen Handling

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood and BAL (bronchoalveolar lavage)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Sample collection — Plasma and BAL sample collection

SUMMARY:
This prospective study will explore the pharmacokinetic exposure and pharmacodynamics of the echinocandins (caspofungin or anidulafungin) in critically ill patients.

DETAILED DESCRIPTION:
This non-randomized, monocenter pharmacokinetic study will be carried out in critically ill patients receiving multiple dose treatment with echinocandins (caspofungin or anidulafungin).

The pharmacokinetics and pharmacodynamics of the echinocandins in plasma and BAL will be determined. Especially, the relative contributions of two pathophysiological alterations (capillary leak and hypoalbuminemia) encountered in critically ill patients, will be explored.

Also other correlating covariates will be identified to provide a rationale for optimal dosing strategy in critically ill patients.

ELIGIBILITY:
Inclusion Criteria:

* Treatment with anidulafungin or caspofungin
* Admitted to an ICU ward

Exclusion Criteria:

* < 18 years
* DNR 2 or 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Critically ill patients.
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2012-09-21 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Area under the curve (AUC) | July 2020
  The area under the concentration-time curve will be calculated
Half-life (T1/2) | July 2020
  The half-life will be calculated
Volume of distribution (Vd) | July 2020
  The volume of distribution will be calculated
Clearance (CL) | July 2020
  The clearance will be calculated
Maximum plasma concentration | July 2020
  The median maximum plasma concentration will be reported
Minimum plasma concentration | July 2020
  The median minimum plasma concentration will be reported
Average plasma concentration | July 2020
  The average plasma concentration will be calculated

SECONDARY OUTCOMES:
Influence of serum creatinin (mg/dL) on echinocandin-exposure | July 2020
Influence of glomerular filtration rate (ml/min) on echinocandin-exposure | July 2020
Influence of on bilirubin on echinocandin-exposure | July 2020
Influence of gamma-GT on echinocandin-exposure | July 2020
Influence of alkaline phosphatase on echinocandin-exposure | July 2020
Influence of AST on echinocandin-exposure | July 2020
Influence of ALT on echinocandin-exposure | July 2020
Influence of SOFA ( sequential organ failure assessment) score on echinocandin-exposure | July 2020
Influence of APACHE II (Acute Physiology and Chronic Health Evaluation II) score on echinocandin-exposure | July 2020
Influence of total protein on echinocandin-exposure | July 2020
Influence of serum albumin on echinocandin-exposure | July 2020
Influence of Ang-1 on echinocandin-exposure | July 2020
Influence of Ang-2 on echinocandin-exposure | July 2020
Influence of VEGF on echinocandin-exposure | July 2020
Influence of inflammation (CRP) on echinocandin-exposure | July 2020
Influence of fluid balance (mL) on echinocandin-exposure | July 2020
Influence of prothrombin time on echinocandin-exposure | July 2020

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Spriet, PharmD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Belgium

IPD SHARING:
Plan to Share IPD: Undecided